CLINICAL TRIAL: NCT05367427
Title: Clinical Trial to Evaluate the Effect of Regular Consumption of a Heath-treated Postbiotic on the Improvement of Symptoms in People With Mild to Moderate Gastrointestinal Disorders Not Associated With Disease
Brief Title: Heat-treated Postbiotic Consumption in Healthy People With Mild to Moderate Gastrointestinal Symptoms
Acronym: BIOPOLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Biopolis S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HULP 6010
Record Dates: First submitted 2022-02-10; First posted 2022-05-10 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-06

CONDITIONS: Healthy; Gastrointestinal Dysfunction

STUDY DESIGN:
Intervention Model Description: Parallel, randomized, double-blind, controlled pilot clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The masking of the study will be achieved through the identical presentation and characteristics of the product to be consumed. The principal investigator will supply the participants with both the experimental product and the placebo, depending on the randomization. Randomization will be done blindly, so that the participants and the researcher will not know which treatment has been assigned (Experimental or Placebo). Six codes have been generated, 3 for each arm (arm 1: 2325, 2329, 2324; arm 2: 2338, 2333, 2331). The unmasking will take place at the end of the experimental period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heat treated postbiotic Bifidobacterium Longum (Experimental): Consumption of 2 capsules/day of Bifidobacterium Longum CECT 7347 (Total daily equivalent of 2.5 x 10^9 CFU)
  Interventions: Dietary Supplement: Heat treated postbiotic Bifidobacterium Longum consumption
- Placebo (Placebo Comparator): Consumption of 2 placebo capsules/day filled with maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Heat treated postbiotic Bifidobacterium Longum consumption — Regular consumption in breakfast of heat treated postbiotic B. longum
  Other Names: Experimental
  Arms: Heat treated postbiotic Bifidobacterium Longum
Dietary Supplement: Placebo — Maltodextrin
  Other Names: Control
  Arms: Placebo

SUMMARY:
The use of probiotics is a widespread clinical practice to improve the composition of the microbiota in healthy and pathological patients. However, in recent years, postbiotics have begun to be used that can exert a certain anti-inflammatory effect at the intestinal level. Among them, Bifidobacterium longum (CECT 7347) has been used in various clinical trials with promising results. It has immunoregulatory properties and an excellent ability to attenuate the activity of epithelial cells at the intestinal level. However, it is necessary to carry out clinical trials to verify its effects, preferably in healthy patients who show certain gastrointestinal discomfort. For this reason, a parallel, randomized, double-blind, controlled pilot clinical trial with 2 study arms has been proposed to assess the effect of habitual consumption of a heat treated postbiotic B. longum CECT 7347 on mild-moderate functional digestive disorders in a group of healthy people.

DETAILED DESCRIPTION:
Recently, there has been a great advance in functional digestive disorders research by new methodological strategies development for their treatment. One of the most interesting line broads the use of microorganisms with the aim of reducing the gastrointestinal. The most studied in this context belong to the genus Bifidobacterium. These microorganisms have shown a remarkable capacity to modulate the inflammatory response, whose efficacy was previously evaluated in celiac patients. Subsequently, different in vitro studies and animal models has been carried out on Bifidobacterium strains, specifically B. longum CECT 7347. Its effect on inflammation caused by gliadins, has reported promising results. This strain is characterized by its anti-inflammatory activity and its ability to recover the intestinal barrier.

Clinical trials in humans took place once the genome of the B. longum CECT 7347 strain and its safety at the level of oral consumption were studied. Continuing with the work carried out in animal models, the efficacy of oral consumption in celiac patients was evaluated, although studies were also carried out on other individuals with liver or dermatological pathologies.

Gastrointestinal symptoms in adults are usually predominant and have important consequences for health and quality of life. In addition, recent studies suggest that the composition of the intestinal microbiota in those people who have gastrointestinal symptoms may come from intestinal dysbiosis, highlighting the role in the noticeable symptoms. Digestive disorders are characterized by compositional imbalances in the gut microbiota, particularly by a reduced number on both total bifidobacteria and Bifidobacterium longum ES1 (CECT 7347). Recent in vitro studies have shown that the presence of B. longum CECT 7347 reduces the toxic and inflammatory effects on intestinal cells.

The former evidences it has been hypothesised that the administration of a heat treated postbiotic B. longum CECT 7347 could modify the composition of the intestinal microbiota due to its immunoregulatory properties and the ability to attenuate the activity of epithelial cells. The proper administrations should attenuate the inflammatory effects, producing a decrease in the prevalence of gastrointestinal symptoms in undiagnosed groups, but which may suffer from a certain intestinal dysbiosis. Based on the above background, a parallel, randomized, double-blind, controlled pilot clinical trial with two study arms has been proposed to assess the effect of habitual consumption of heat treated postbiotic B. longum CECT 7347 on mild to moderate functional digestive disorders in a group of healthy people.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who obtain a score between 13 and 39 points with diarrhea predominance in the Gastrointestinal Symptoms Rating Scale (GSRS-IBS) corresponding to the last week.
* Men and women between 18 and 65 years old.
* Absence of a family or social environment that prevents compliance with treatment.
* Adequate cultural level and understanding of the clinical study.
* Agree to voluntarily participate in the study and give their informed consent in writing.

Exclusion Criteria:

* Subjects with BMI <18.5 or >35 kg/m2.
* Subjects who have participated in programs and/or clinical trials and who have lost or gained more than 4 kg in the last 3 months.
* Subjects diagnosed with Diabetes Mellitus 1 or 2.
* Subjects diagnosed with metabolic syndrome, hypothyroidism and/or hyperthyroidism.
* Subjects with allergies to the excipients of the product/placebo.
* Subjects with an established diagnosis of eating behavior disorder.
* Women who do not agree to continue with their contraceptive method during the study period.
* Subjects who perform excessive physical exercise (>2 h more than 3 times per week).
* Subjects who wish to start an exercise plan and/or dietary program during the study period.
* Subjects with serious diseases (liver disease, kidney disease, heart disease, lung disease, cancer, etc.).
* Subjects with chronic intestinal pathologies (gastritis, ulcerative colitis, irritable bowel syndrome, inflammatory bowel disease, Crohn's disease, intestinal perforation, history of gastroparesis, etc.).
* Subjects with autoimmune diseases and/or subjects undergoing treatment with corticosteroids, immunosuppressants and/or biologicals in the last 12 months.
* Subjects with major surgeries in the last 3 months or gastrointestinal surgery in the last 6 months.
* Subjects with weight loss surgery (gastric bypass, lap band)
* Subjects under treatment with oral antibiotics during the 30 days prior to the start of the study.
* Subjects with recent episodes of acute gastrointestinal illness such as nausea, vomiting or acute gastroenteritis 2 weeks before the start of the study.
* Subjects who wish to quit smoking during the duration of the study.
* Subjects who consume antioxidant supplements, omega 3 supplements, vitamins, minerals, prebiotic, synbiotic, parabiotic or probiotic products in the 4 weeks prior to the start of the study and who do not agree to suppress their consumption during the study period.
* Subjects with alcohol consumption greater than 30 g/day (equivalent to 300 ml of wine, about 3 beers or a glass (75 ml) of whisky, cognac, anise, etc.)).
* Subjects with regular use of antidiarrheal medications (>2 per week) during the last 3 months prior to the start of the study.
* Subjects on anticoagulant therapy.
* Subjects with dementia, mental illness, or decreased cognitive function.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of gastrointestinal symptoms | Day 0 - Day 60
  Changes in the score obtained through the Gastrointestinal Symptom Rating of Irritable Bowel Syndrome (GSRS-IBS) scale (Score range: 0-78 points). A greater score means a higher occurrence of gastrointestinal symptoms.

SECONDARY OUTCOMES:
Frequency of gastrointestinal symptoms | Day 0 - Day 60
  Changes in the score obtained through the Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) scale (Score range: 0-500 points). A greater score punctuation means a higher frequency of gastrointestinal symptoms.
Gastrointestinal quality of life | Day 0 - Day 60
  Changes in the score obtained in the gastrointestinal quality of life questionnaire (GIQLI) (Score range: 0-144 points). A higher score means a better perception of gastrointestinal quality of life.
Defecation pattern | Day 0-Day 60
  Modifications in the defecation pattern of the Bristol Scale, decreasing stools with a 5-7 assessment and observing a greater presence of stools with a 3-4 value. Ideal scores range between 3-4; constipation occurs in 1-2 scores and the presence of diarrhoea in highlighted with stools of 5, 6 and 7 description.
Visceral sensitivity | Day 0- Day 60
  Changes in Visceral Sensitivity Index (VSI) score (Range: 15-90). A lower score means an undesirable visceral sensitivity.
Zonulin concentration | Day 0 - Day 60
  Changes in fecal zonulin concentration, as a biomarker related to increased intestinal permeability
Faecal microbiome analysis | Day 0 vs Day 60
  Changes in feacal microbiome after heat treated postbiotic
Glucose | Day 0 - Day 60
  Maintenance of biochemical parameters within normal concentrations (74-106 mg/dL)
Total serum protein | Day 0 - Day 60
  Maintenance of biochemical parameters within normal concentrations of total serum proteins (range from 6.4 to 8.3 g/dL)
Serum albumin | Day 0 - Day 60
  Maintenance of biochemical parameters within normal concentrations of serum albumin (range from 3.4 to 5.4 g/dL)
HDL-cholesterol | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of HDL-cholesterol (♂: >40, ♀: >50 mg/dL)
Serum prealbumin | Day 0 - Day 60
  Maintenance of biochemical parameters within normal concentrations of serum prealbumin (range from 17 to 42 mg/dL)
Cholesterol | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of total cholesterol (<200 mg/dL)
LDL-cholesterol | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of LDL-cholesterol (<130 mg/dL)
Triglycerides | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of triglycerides (TG) (<150 mg/dL)
Vitamin A | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of vitamin A (0.3-0.7 ug/mL)
Vitamin E | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of vitamin E (5-20 ug/mL)
Vitamin D | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of vitamin D (30-100 ng/mL)
Calcium | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of Calcium (8.6-10,2 mg/dL)
Phosphorus | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of Phosphorus (2.5-4.5 mg/dL)
Sodium | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of Sodium (136-145 mmol/L)
Potassium | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of Potassium (3.5-5.1 mmol/L)
Magnesium | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of Magnesium (1.60-2.60 mg/dL)
Chlorine | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of Chlorine (99-109 mmol/L)
Folic Acid | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of Folic Acid (>2,6 ng/dL)
Vitamin B12 | Day 0 - Day 60
  Maintenance of biochemical parameters within normal serum concentrations of Vitamin B12 (211-911 pg/mL).
Interleukins | Day 0 - Day 60
  Changes in inflammatory m. These biomarkers are measured in pg/mL
C-reactive protein (CRP) | Day 0 - Day 60
  Modifications in the C-reactive protein (CRP). This biomarker is measured in mg/L
Body weight | Day 0 - Day 60
  Changes produced in body weight measured in kilograms
Waist circumference | Day 0 - Day 60
  Data referring to the waist circumference of the Spanish population allow to estimate cardiovascular risk parameters from 95 cm in men and 82 cm in women, and very high risk from 102 cm in men and 90 cm in women. The measurement is taken at the narrowest point between the last rib and the iliac crest, with the tape against the skin but not compressed. The person should be kept in an upright position, distributing the weight equally on both legs and their arms relaxed at the sides of the body.
Body mass index (BMI) | Day 0 - Day 60
  Relationship between body weight (kg) and height (m) squared of the individual: Weight/(Height)2
Fat mass percentage | Day 0 - Day 60
  Changes or maintenance of the fat mass % measured by electrical bioimpedance
Muscle Mass percentage | Day 0 - Day 60
  Changes or maintenance of the muscle mass % measured by electrical bioimpedance
Blood pressure | Day 0 - Day 60
  Maintenance in systolic pressure and diastolic pressure measured by blood pressure monitor
Heart rate | Day 0 - Day 60
  Heart rate maintenance measured in beats per minute (bpm) using blood pressure monitor
Tolerance | Day 0 - Day 60
  Changes measured by applying a tolerance questionnaire that evaluates qualitative information on possible symptoms associated with the consumption of the product such as: nausea, heartburn, diarrhea, abdominal distension or halitosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Health Research IdiPAZ, Madrid, Spain